CLINICAL TRIAL: NCT00913913
Title: A Phase II Study of VEGF Blockade With Bevacizumab Combined With Autologous Tumor/Dendritic Cell Vaccine (DC Vaccine), Interleukin-2 (IL-2) and Interferon-α-2b (IFNα-2b) in Patients With Metastatic Renal Cell Carcinoma (RCC)
Brief Title: Bevacizumab, Autologous Tumor/DC Vaccine, IL-2 and IFNα-2b in Metastatic Renal Cell Carcinoma (RCC) Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual not allowing site to meeting statistical endpoints
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0708; R01CA095648 (NIH)
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Results first posted 2015-12-01 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2014-02

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — lentiviral minigene vaccine of COVID-19 coronavirus; Bevacizumab; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bevacizumab,IL-2, IFN, DC vaccine (Experimental): Patients will be dosed with bevacizumab (10mg/kg) intravenously every two weeks beginning four weeks prior to the first vaccine. Each treatment week includes ultrasound guided intranodal DC-vaccine injection (1 X 107 cells/1mL), followed by 5 days of continuous intravenous infusion of IL-2 (18 MiU/m2), and three subcutaneous injections of IFNa-2b (6 MiU) (every other day)
  Interventions: Biological: DC vaccine; Drug: Bevacizumab; Biological: IL-2; Biological: IFN

INTERVENTIONS:
Biological: DC vaccine — DC Vaccine therapy 10E7 intranodally every cycle
Drug: Bevacizumab — Bevacizumab 10mg/kg iv every 2 weeks
  Other Names: Avastin
Biological: IL-2 — IL-2 18 MiU/m2 CI 5 days
Biological: IFN — IFN 6 MiU subc TIW

SUMMARY:
Immune therapies, such as a IL-2, for metastatic renal cell carcinoma (mRCC) are designed to mobilize immune effector cells that recognize and destroy cancer. The investigators have recently observed a 50% objective response rate (16% CR) in mRCC patients treated with autologous tumor lysate -dendritic cell (DC)-vaccine, IL-2 and interferon alfa (IFN). New agents inhibiting vascular endothelial growth factor (VEGF) pathways have demonstrated significant benefit in mRCC patients as well, but rarely induce CRs. High blood VEGF is associated with poor response to IL-2 and can cause tumor specific immune dysregulation. To test whether complementary mechanisms of immune activation and disruption of regulatory pathways enhance outcome the investigators plan to treat 24 mRCC patients in a phase II trial using bevacizumab, DC vaccine, IL-2, and IFN. Observations from this project will be used in the development of novel cancer therapies which, if successful, will decrease the burden of cancer on the public.

The investigators propose to determine 1) the objective clinical response rate to treatment and progression free survival, 2) the clinical and autoimmune related toxicity profile of therapy, and 3) the treatment related tumor-specific immune response and the relationship of tumor-specific immune response and objective clinical response.

DETAILED DESCRIPTION:
All eligible patients will receive a total of five treatment weeks, each consisting of approximately 5 days. Prior to therapy, patients will undergo apheresis for DC preparation. DC-Tumor vaccines will be frozen in 90% pooled human AB serum/ 10% DMSO to be used for treatment Patients will be dosed with bevacizumab (10mg/kg, Genentech) intravenously every two weeks beginning four weeks prior to the first vaccine. Each treatment week includes ultrasound guided intranodal DC-vaccine injection (1 X 107 cells/1mL), followed by 5 days of continuous intravenous infusion of IL-2 (18 MiU/m2, Novartis), and three subcutaneous injections of IFNa-2b (6 MiU, Schering -Plough Corp.) (every other day). The first two treatment weeks, the induction phase, will be separated by a 9 day rest. Three additional treatment weeks, the maintenance phase, will be separated by 23 rest days.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic renal cell carcinoma with measurable disease.
2. Adequate tumor tissue properly stored and available to produce lysate for a minimum of three vaccine preparations.
3. Patients must be at least 4 weeks from their last therapy (tyrosine kinase inhibitors, immunotherapy, radiation, surgery or chemotherapy (6 weeks for nitrosureas) and recovered from all ill effects.
4. Have measurable disease.
5. Patients must be at least 4 weeks from major surgery, 1 week from minor surgery, and recovered from all ill effects.
6. Karnofsky Performance Status ≥80%.
7. Adequate end organ function:
8. Women should not be lactating and, if of childbearing age, have a negative pregnancy test within two weeks of entry to the study.
9. Appropriate contraception in both genders.
10. The patient must be competent and have signed informed consent.
11. Patients may have received one prior therapy with targeted therapies (e.g. sorafenib and sunitinib).

Exclusion Criteria:

1. Patients who have previously received bevacizumab or IL-2 are not eligible.
2. Concomitant second malignancy except for non-melanoma skin cancer, and non-invasive cancer such as cervical CIS, superficial bladder cancer without local recurrence or breast CIS.
3. In patients with a prior history of invasive malignancy, less than five years in complete remission.
4. Positive serology for HIV, hepatitis B or hepatitis C which should be confirmed with antigenemia.
5. Significant co-morbid illness such as uncontrolled diabetes or active infection that would preclude treatment on this regimen.
6. Use of corticosteroids or other immunosuppression (if patient had been taking steroids, at least 2 weeks must have passed since the last dose). Inhaled steroids > 1000mcg beclomethasone per day or its equivalent.
7. History of inflammatory bowel disease or other serious autoimmune disease. (Not including thyroiditis and rheumatoid arthritis).
8. Patients with organ allografts.
9. Uncontrolled hypertension (BP >150/100 mmHg).
10. Proteinuria dipstick > 3+ or > 2gm/24 hours, or a urine protein:creatinine ratio > 1.0 at screening.
11. Major surgery, open biopsy, significant traumatic injury within 28 days of starting treatment or anticipation of need for major surgical procedure during the course of the study.
12. Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to starting treatment. Central venous catheter placements are permitted.
13. History of abdominal fistula, gastrointestinal perforation, or intrabdominal abscess within 6 months prior to starting treatment.
14. Serious, non-healing wound, ulcer, or bone fracture.
15. History of tumor-related or other serious hemorrhage, bleeding diathesis, or underlying coagulopathy.
16. History of deep venous thrombosis, or other thrombotic event within the past six months or clinically significant peripheral vascular disease.
17. Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc S Ernstoff, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Background] Ernstoff MS, Crocenzi TS, Seigne JD, Crosby NA, Cole BF, Fisher JL, Uhlenhake JC, Mellinger D, Foster C, Farnham CJ, Mackay K, Szczepiorkowski ZM, Webber SM, Schned AR, Harris RD, Barth RJ Jr, Heaney JA, Noelle RJ. Developing a rational tumor vaccine therapy for renal cell carcinoma: immune yin and yang. Clin Cancer Res. 2007 Jan 15;13(2 Pt 2):733s-740s. doi: 10.1158/1078-0432.CCR-06-2064. PMID 17255302

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab,IL-2, IFN, DC Vaccine
Started | 8
Completed | 0
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: Number was the actual number of patients who signed consent and received treatment on study.
Arm/Group | Bevacizumab,IL-2, IFN, DC Vaccine
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] — Age is the mean of the age of the 8 patients at time of consent for study participation.
  years | 55 [50 to 70]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: median progression free survival
Time Frame: 5 years
Measure: Median (Full Range); unit: DAYS
Arm/Group | Bevacizumab,IL-2, IFN, DC Vaccine
Number analyzed (Participants) | 8
DAYS | 340 [73 to 1582]

2. Secondary Outcome: To Characterize the Number of Participants With Clinical and Autoimune Related Toxicity of Treatment
Description: To characterize the clinical and autoimmune related toxicity profile of the combined treatment regimen using CTCAE 3. Toxicity reported are those expected from high dose IL-2 and were not considered adverse events.
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Bevacizumab,IL-2, IFN, DC Vaccine
Number analyzed (Participants) | 8
participants | 8

3. Other Pre Specified Outcome: Measure of Percent of CD4 and CD8 Lymphocyte Subsets
Description: percent of CD4 and CD8 positive lymphocyte subsets
Time Frame: Baseline, day 28, day 70
Population: Peripheral blood lymphocyte subsets: 5 subjects at baseline and same 5 at day 70. 6 subjects analyzed at day 28
Measure: Mean (Full Range); unit: percentage of total lymphocytes
Arm/Group | Bevacizumab,IL-2, IFN, DC Vaccine
Number analyzed (Participants) | 6
percentage of total lymphocytes
  CD4 Central memory: baseline | 0.50 [0.21 to 1.42]
  CD4 Central memory: Day 28 | 1.71 [0.80 to 2.60]
  CD4 Central memory: Day 70 | 0.69 [0.14 to 1.93]
  CD8 Central memory: baseline | 1.61 [0.32 to 5.36]
  CD8 Central memory: day 28 | 4.74 [2.49 to 7.79]
  CD8 Central memory: day 70 | 2.76 [0.18 to 9.84]

4. Other Pre Specified Outcome: Clinical Response
Description: clinical response by RECIST 1.1
Time Frame: Day 70
Measure: Number; unit: participants
Arm/Group | Bevacizumab,IL-2, IFN, DC Vaccine
Number analyzed (Participants) | 8
participants | 4

ADVERSE EVENTS:
Time Frame: From time patient first dosed with any study specific medications to end of study. Subjects were evaluated until progression. The median time of follow up was 340 days with a range from 73 to 1582 days.
Arm/Group | Bevacizumab,IL-2, IFN, DC Vaccine
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab,IL-2, IFN, DC Vaccine (N=8)
hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) — grade 4 hepatobiliary dysfunction related to IL-2 therapy
Liver dysfunction/Failure (Hepatobiliary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study closed early due to difficulty enrolling patients with enrollment limited due to new competing therapies. Though enrollment numbers per statistical design were not met, the primary objective may still be reviewed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes